CLINICAL TRIAL: NCT02174250
Title: Effect of a Strong Enzyme Inducer, Rifampin, on the Single-Dose Pharmacokinetics of Istradefylline in Healthy Subjects
Brief Title: The Effect of Rifampin on the Metabolism of Istradefylline in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 6002-015
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease
Keywords: PD
MeSH Terms: conditions — Parkinson Disease | interventions — istradefylline; Rifampin; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Istradefylline 40mg (Experimental): Period 1: Day 1, istradefylline 40mg then crossover to Period 2
  Interventions: Drug: Istradefylline 40 mg
- Rifampin 300mg BID + istradefylline 40mg (Experimental): Period 2: Days 1-20 rifampin 300mg BID + istradefylline 40mg Day 8 only
  Interventions: Drug: Istradefylline 40 mg; Drug: Rifampin 300mg BID + istradefylline 40mg Day 8 only

INTERVENTIONS:
Drug: Istradefylline 40 mg — On Day 1, istradefylline 1 × 40-mg tablet administered alone
  Other Names: KW-6002
Drug: Rifampin 300mg BID + istradefylline 40mg Day 8 only — On Days 1 - 20, rifampin 300mg BID; On Day 8, istradefylline 40 mg administered first with rifampin about 2 hours after istradefylline administration
  Other Names: rifadin
  Arms: Rifampin 300mg BID + istradefylline 40mg

SUMMARY:
The purpose of this study is to test whether Rifampin affects blood levels of istradefylline in humans. Rifampin could possibly decrease istradefylline levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking male and post-menopausal female subjects
* Body Mass Index: 18.0-35.0 kg/m2, inclusive
* Subjects must not be taking drugs that are moderate to potent inhibitors of CYP3A4 or CYP1A2.
* Subjects without clinically significant medical history in the judgment of the investigator
* Subjects without clinically significant laboratory or ECG abnormalities

Exclusion Criteria:

* Females that are pregnant or lactating
* Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study;
* Known history of treatment for drug or alcohol addiction within the previous 12 months;
* Subjects with an average alcohol intake of more than 2 units per day or 14 units per week up to 48 hours prior to the istradefylline dose on Day 1. One unit of alcohol is ½ pint of beer (285 mL) or 1 glass of spirits (25 mL) or 1 glass of wine (125 mL);
* Donated or lost > 500 mL of blood within 3 months prior to istradefylline dose on Day 1 of Period 1;
* Positive test results for human immunodeficiency virus (HIV) or Hepatitis B surface antigen, or Hepatitis C;
* Positive test results for drugs of abuse at screening;
* Unable, or unwilling to tolerate multiple venipunctures;
* Difficulty fasting or eating the standard meals that will be provided;
* Use of tobacco or nicotine-containing products within 90 days of the study start to the Follow-up visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to infinity (AUC0 ∞) and Observed maximum plasma concentration (Cmax) of istradefylline | Intermittently for a total of 62 days

SECONDARY OUTCOMES:
Number of serious adverse events, and non-serious adverse events | Continuously for up to 74 days

CONTACTS AND LOCATIONS:
Overall Officials: Marc Cantillon, M.D., Study Chair — Kyowa Hakko Kirin Pharma, Inc.; Amy Zhang, PhD, Study Director — Kyowa Hakko Kirin Pharma, Inc.
Locations (1):
- Celerion, Inc., Tempe, Arizona, United States